CLINICAL TRIAL: NCT00762983
Title: Claritin® Tablet 10 mg, Claritin® RediTabs® 10 mg, Claritin® Dry Syrup 1% Drug Use Investigation (Pediatrics)
Brief Title: Observation of Use of Claritin (Loratadine) Tablet, RediTabs, and Dry Syrup in Children (Study P05834)(COMPLETED)
Status: Completed | Type: Observational
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: P05834
Record Dates: First submitted 2008-09-29; First posted 2008-09-30 (Estimated); Last update posted 2015-02-13 (Estimated); Status verified 2015-02

CONDITIONS: Rhinitis, Allergic, Seasonal; Rhinitis, Allergic, Perennial; Urticaria; Pruritus
MeSH Terms: conditions — Rhinitis, Allergic, Seasonal; Rhinitis, Allergic, Perennial; Urticaria; Pruritus | interventions — Loratadine

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Group 1: Pediatric patients who are treated with Claritin for any of the following reasons: allergic rhinitis, urticaria, itching due to skin disease (eczema, dermatitis, or pruritus cutaneous)
  Interventions: Drug: loratadine

INTERVENTIONS:
Drug: loratadine — Claritin Tablet 10 mg, Claritin RediTabs 10 mg: For pediatric patients aged 7 years and older, 10 mg of loratadine is orally administered once daily after a meal in usual cases.
  Claritin Dry Syrup 1%: For pediatric patients aged 3 to < 7 years, 5 mg loratadine (0.5 g dry syrup); and for pediatric patients aged 7 years and older, 10 mg of loratadine (1 g dry syrup) is dissolved immediately before use and orally administered once daily after a meal in usual cases.
  The observation period will not be specified.
  Other Names: Claritin, SCH 29851

SUMMARY:
The purpose of this study is to collect information on unexpected adverse reactions (ADRs), how often ADRs occur, and factors that can affect the safety and effectiveness of Claritin (loratadine) when used in children. Patients will be observed while they are taking Claritin, and ADRs and symptom scores will be recorded. At the end of treatment, improvement in symptoms will be recorded.

Post-marketing surveys are not considered applicable clinical trials and thus the results of this survey will not be posted at its conclusion. The results will be submitted to public health officials as required by applicable national and international laws.

ELIGIBILITY:
Inclusion Criteria:

* Pediatric patients aged 3 to 15 years who are treated with Claritin for any of the following reasons: allergic rhinitis, urticaria, itching due to skin disease (eczema, dermatitis, or pruritus cutaneous)

Exclusion Criteria:

* (None)

Ages: 3 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Pediatric patients who are treated with Claritin at a department of pediatrics, department of otorhinology, department of dermatology, etc. at approximately 120 institutions
Sampling Method: Non-Probability Sample
Enrollment: 1003 (Actual)
Dates: Start 2008-03; Primary Completion 2009-02 (Actual); Study Completion 2009-02 (Actual)

PRIMARY OUTCOMES:
Unexpected adverse drug reactions (ADRs) that had not been detected in pre-approval clinical studies | During and at the end of the observation period
Allergic rhinitis: nasal symptom scores (paroxysmal sneeze, nasal discharge, nasal congestion, and intranasal itching) | Before the start of treatment, during the observation period, and at the end of the observation period
Urticaria, eczema, dermatitis, pruritus cutaneous: severity score of itching | Before the start of treatment, during the observation period, and at the end of the observation period

SECONDARY OUTCOMES:
Allergic rhinitis: Markedly improved, Moderately improved, Mildly improved, Unchanged, Worsened, Unassessable | At the end of the observation period
Urticaria, eczema, dermatitis, pruritus cutaneous: Resolved, Improved, Unchanged, Worsened, Unassessable | At the end of the observation period